CLINICAL TRIAL: NCT04726345
Title: Effect of Antihistamines on Ureteral Stent-Related Symptoms: Randomized Controlled Trial
Brief Title: Effect of Antihistamines on Ureteral Stent-Related Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Coloplast A/S (Industry)
Responsible Party: Principal Investigator, Ojas Shah, George F. Cahill Professor of Urology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AAAT0219
Record Dates: First submitted 2021-01-20; First posted 2021-01-27 (Actual); Results first posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Nephrolithiasis
Keywords: Antihistamines; Ureteral stent
MeSH Terms: conditions — Nephrolithiasis | interventions — fexofenadine

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1 ratio to receive fexofenadine or placebo in addition to the standard of care. A total of 39 subjects will be randomized to each group.
Who Masked: Participant, Care Provider
Masking Description: Subjects and the study urologist will be blinded to treatment allocation. Treatment allocation will be known by the investigator performing data analysis, who will not be directly participating in patient care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fexofenadine (Experimental): Participants in this arm will receive fexofenadine 180mg once daily, in addition to standard of care pain medications (NSAIDs).
  Interventions: Drug: Fexofenadine Hcl 180Mg Tab
- Placebo (Placebo Comparator): Participants in this arm will receive placebo once daily, in addition to standard of care pain medications (NSAIDs).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fexofenadine Hcl 180Mg Tab — Fexofenadine 180mg tablet to be taken orally once a day until stent removal.
  Other Names: Fexofenadine
  Arms: Fexofenadine
Drug: Placebo — Placebo tablet to be taken orally once a day until stent removal.
  Other Names: Placebo Tablet
  Arms: Placebo

SUMMARY:
This is a prospective, double-blind, randomized, open-label, single-center trial of up to 78 participants who are adult patients (aged 18-80 years) and are undergoing unilateral retrograde ureteroscopy with planned ureteral stent placement for treatment of urinary tract stones. Eligible patients will be randomly and divided into two groups in a 1:1 ratio. Group A will receive fexofenadine 180 mg once daily in addition to standard of care treatment. Group B will receive placebo in addition to standard of care treatment. The routine standard of care treatment will consist of oral non-steroidal anti-inflammatory drugs (NSAIDs).

The primary outcomes of the study are the Ureteral Stent Symptom Questionnaire (USSQ) urinary symptom score and pain score. Secondary outcomes include (i) number of office phone calls due to urinary symptoms; (ii) duration of analgesic use; (iii) duration and quantity of narcotic use; (iv) number of emergency department visits; (v) drug-related adverse effects; (vi) other domains of the USSQ.

DETAILED DESCRIPTION:
Ureteral stents treat ureteral obstruction, allow for passive dilation of the ureter, maintain urine flow to the bladder, and aid in the recovery of the ureter after endoscopic surgery or ureteral injury. These stents are routinely utilized after urologic procedures for the treatment of urolithiasis and are generally kept in place for 1-2 weeks following the procedure. Despite their advantages, indwelling ureteral stents cause discomfort and reduce patient quality of life. These symptoms are partially attributed to local irritation to the ureter and bladder. Bothersome stent-related symptoms include urinary urgency, frequency, flank pain, hematuria, dysuria, sexual side effects, and emotional distress. The majority of patients with ureteral stents experience symptoms post-operatively.

Several studies have indicated that agents such as antimuscarinics or alpha-1 adrenergic receptor antagonists may improve stent-related symptoms. The indications for anticholinergic medications are based on blocking involuntary bladder muscle contraction; however, the efficacy of these drugs is still controversial. Furthermore, these medications have potential adverse side effects.

Antihistamines also show potential in alleviating stent-related symptoms. Multiple in vitro studies have shown H1 receptor activity involved both in ureteral peristalsis and in bladder contraction. Both first- and second-generation H1 antagonists have shown activity in the urinary tract. In clinical practice, antihistamines are commonly utilized in the management of bladder pain caused by interstitial cystitis. Additionally, a randomized controlled trial found efficacy of antihistamines for pain management in the setting of renal colic from obstructing ureteral stones. There is novel evidence that in patients with indwelling stents, there are inflammatory changes in the bladder with an associated eosinophilic reaction. Eosinophilic cystitis is commonly associated with bladder irritation or allergy, and these findings point to a novel paradigm of treating patients with antihistamines. To our knowledge, no studies have evaluated the efficacy of antihistamines for managing stent-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18-80 years) who are undergoing unilateral retrograde ureteroscopy with planned ureteral stent placement for treatment of urinary tract stones

Exclusion Criteria:

* Preoperative use of antihistamines, beta-3 agonists, anticholinergics, corticosteroids, and chronic opioid analgesic use
* Preoperative indwelling ureteral stent at the time of treatment
* Neurogenic bladder, ureteral stricture, interstitial cystitis, or chronic prostatitis
* Pregnancy or breastfeeding
* Planned bilateral ureteroscopy
* Solitary or transplanted kidney
* Hypersensitivity to antihistamines
* Severe renal disease (glomerular filtration rate (GFR) < 10 ml/min or on dialysis)
* Significant deviation in operative plan (ureteral stent not deemed necessary, incidental urologic malignancy, tandem ureteral stent placement, second-stage procedure required)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ojas Shah, MD, Principal Investigator — Professor of Urology
Locations (1):
- Columbia University Irving Medical Center/NYP, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aboutaleb H, Gawish M. Correlation of Bladder Histopathologic Changes Due to Double-J Stenting to the Period of Stenting: A Preliminary Study. J Endourol. 2017 Jul;31(7):705-710. doi: 10.1089/end.2017.0113. Epub 2017 May 31. PMID 28467731
- [Background] Joshi HB, Newns N, Stainthorpe A, MacDonagh RP, Keeley FX Jr, Timoney AG. Ureteral stent symptom questionnaire: development and validation of a multidimensional quality of life measure. J Urol. 2003 Mar;169(3):1060-4. doi: 10.1097/01.ju.0000049198.53424.1d. PMID 12576846
- [Background] Joshi HB, Stainthorpe A, MacDonagh RP, Keeley FX Jr, Timoney AG, Barry MJ. Indwelling ureteral stents: evaluation of symptoms, quality of life and utility. J Urol. 2003 Mar;169(3):1065-9; discussion 1069. doi: 10.1097/01.ju.0000048980.33855.90. PMID 12576847
- [Background] Lamb AD, Vowler SL, Johnston R, Dunn N, Wiseman OJ. Meta-analysis showing the beneficial effect of alpha-blockers on ureteric stent discomfort. BJU Int. 2011 Dec;108(11):1894-902. doi: 10.1111/j.1464-410X.2011.10170.x. Epub 2011 Mar 31. PMID 21453351
- [Background] Lingeman JE, Preminger GM, Goldfischer ER, Krambeck AE; Comfort Study Team. Assessing the impact of ureteral stent design on patient comfort. J Urol. 2009 Jun;181(6):2581-7. doi: 10.1016/j.juro.2009.02.019. Epub 2009 Apr 16. PMID 19375088
- [Background] Sivalingam S, Streeper NM, Sehgal PD, Sninsky BC, Best SL, Nakada SY. Does Combination Therapy with Tamsulosin and Tolterodine Improve Ureteral Stent Discomfort Compared with Tamsulosin Alone? A Double-Blind, Randomized, Controlled Trial. J Urol. 2016 Feb;195(2):385-90. doi: 10.1016/j.juro.2015.08.104. Epub 2015 Sep 21. PMID 26393904
- [Background] Yilmaz E, Batislam E, Deniz T, Yuvanc E. Histamine 1 receptor antagonist in symptomatic treatment of renal colic accompanied by nausea: two birds with one stone? Urology. 2009 Jan;73(1):32-6. doi: 10.1016/j.urology.2008.08.494. Epub 2008 Oct 11. PMID 18849063
- [Derived] Han DS, Margolin EJ, Movassaghi M, Johnson JP, Chowdhury M, Pingle SR, Schulster ML, Weiner DM, Shah O. Effect of Antihistamine on Ureteral Stent-Related Symptoms: A Double-Blind Randomized Controlled Trial. Urol Pract. 2025 Jul;12(4):415-425. doi: 10.1097/UPJ.0000000000000791. Epub 2025 Feb 12. PMID 39937815

RESULTS

PARTICIPANT FLOW:
Period: Baseline Analysis
Arm/Group | Fexofenadine | Placebo
Started | 39 | 39
Completed | 37 | 36
Not Completed | 2 | 3
Period: Stent in Situ
Arm/Group | Fexofenadine | Placebo
Started | 37 | 36
Completed | 35 | 36
Not Completed | 2 | 0
Period: Post-stent Removal Follow-up (4-6 Weeks)
Arm/Group | Fexofenadine | Placebo
Started | 35 | 36
Completed | 34 | 35
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: Of the 78 participants who enrolled in the study, 5 withdrew prior to baseline data collection.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fexofenadine | Placebo | Total
Number analyzed (Participants) | 37 | 36 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (11) | 52 (15) | 53 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 23 | 21 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 13 | 31
  Not Hispanic or Latino | 19 | 23 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 15 | 20 | 35
  Black | 3 | 3 | 6
  Hispanic or Latino | 18 | 13 | 31
  Asian | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 36 | 73

OUTCOME MEASURES:

1. Primary Outcome: USSQ Urinary Symptom Score
Description: Ureteric Stent Symptoms Questionnaire (USSQ) is a self-administered questionnaire to evaluate the overall impact of ureteral stents on different aspects of life. Urinary symptom will be assessed at different time points. The urinary symptom section consists of 11 questions. The total score range is 11 to 54 points. Higher scores represent increasing symptom severity.
Time Frame: Baseline, stent in situ immediately before stent removal, and poststent removal (4 to 6-week follow-up)
Population: 2 participants (1 in each Arm) were lost to follow-up
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Fexofenadine | Placebo
Number analyzed (Participants) | 35 | 36
score on a scale
  stent in situ | 28 [26 to 31] | 29 [26 to 31]
  follow-up: number analyzed (Participants) | 34 | 35
  follow-up | 16 [15 to 18] | 17 [15 to 18]

2. Primary Outcome: USSQ Body Pain Score
Description: Ureteric Stent Symptoms Questionnaire (USSQ) is a self-administered questionnaire to evaluate the overall impact of ureteral stents on different aspects of life. Body pain will be assessed at different time points. The body pain section consists of 7 questions. The total score range is 0 to 37 points. Higher scores represent increasing pain.
Time Frame: Baseline, stent in situ immediately before stent removal, and poststent removal (4 to 6-week follow-up)
Population: 2 participants (1 in each Arm) were lost to follow-up
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Fexofenadine | Placebo
Number analyzed (Participants) | 35 | 36
score on a scale
  baseline | 11 [7 to 14] | 11 [8 to 15]
  stent in situ | 14 [10 to 18] | 17 [13 to 21]
  follow-up: number analyzed (Participants) | 34 | 35
  follow-up | 2 [0 to 4] | 4 [1 to 6]

3. Secondary Outcome: Number of Office Phone Calls Due to Urinary Symptoms and Pain
Description: This is to measure the morbidity associated with the indwelling ureteral stent. Urinary symptoms will include urinary frequency, urgency, incontinence, nocturia, incomplete emptying, dysuria, and hematuria. Total number of calls per group are reported.
Time Frame: After stent removal (1-2 weeks after surgery)
Measure: Number; unit: office phone calls
Arm/Group | Fexofenadine | Placebo
Number analyzed (Participants) | 37 | 36
office phone calls | 5 | 9

4. Secondary Outcome: Duration of NSAID Use
Description: This is to measure morbidity associated with the indwelling ureteral stent. Duration will be reported in days.
Time Frame: After stent removal (1-2 weeks after surgery)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fexofenadine | Placebo
Number analyzed (Participants) | 37 | 36
days | 3 (3) | 3 (3)

5. Secondary Outcome: Quantity of Narcotic Use
Description: This is to measure the morbidity associated with the indwelling ureteral stent. It will be reported in milligram morphine equivalents.
Time Frame: After stent removal (1-2 weeks after surgery)
Measure: Mean (Standard Deviation); unit: milligram morphine equivalents
Arm/Group | Fexofenadine | Placebo
Number analyzed (Participants) | 37 | 36
milligram morphine equivalents | 1 (5) | 9 (50)

6. Secondary Outcome: Number of Emergency Department Visits
Description: This is to measure morbidity associated with the indwelling ureteral stent. Incidence will be collected at study visit.
Time Frame: After stent removal (1-2 weeks after surgery)
Measure: Number; unit: emergency department visits
Arm/Group | Fexofenadine | Placebo
Number analyzed (Participants) | 37 | 36
emergency department visits | 2 | 3

7. Secondary Outcome: Number of Drug-related Adverse Effects
Description: This is to measure the morbidity of the study drug. Incidence will be self-reported by patients.
Time Frame: After stent removal (1-2 weeks after surgery)
Measure: Number; unit: drug-related adverse effect
Arm/Group | Fexofenadine | Placebo
Number analyzed (Participants) | 37 | 36
drug-related adverse effect | 1 | 0

ADVERSE EVENTS:
Time Frame: Postoperatively, 1-2 weeks after surgery
Arm/Group | Fexofenadine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/36
Other Adverse Events (participants affected / at risk) | 2/37 | 0/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fexofenadine (N=37) | Placebo (N=36)
Dizziness (General disorders) | 1 | 0
UTI (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT04726345/Prot_SAP_000.pdf